CLINICAL TRIAL: NCT06927778
Title: Effects of Corrective Exercises on Trunk Endurance, Jumping Performance and Reaction Time in Adolescent Fencers
Brief Title: Effects of Corrective Exercises in Adolescent Fencers
Acronym: FMS exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Seda Uluşahin, Principal Investigator, Pt PhD, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-227
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Postural Imbalance; Muscle Weakness; Athletic Performance
Keywords: Postural Balance; Adolescent Athletes; Fencing; Core Stability
MeSH Terms: conditions — Muscle Weakness | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Exercise
- No Intervention (No Intervention)

INTERVENTIONS:
Other: Exercise — Individualised corrective exercise protocols based on Functional Movement Screening
  Arms: Intervention

SUMMARY:
The goal is to learn if a Functional Corrective Training (FCT) exercise program improves posture, core muscle endurance, jumping ability, and reaction time in adolescent fencers.

The main questions it aims to answer are:

Does the FCT program improve trunk muscle endurance?

Does the FCT program enhance athletic performance, such as jump height and reaction time?

Researchers will compare adolescent fencers who receive an 8-week FCT exercise program to those who continue regular training only.

Participants will:

Be assigned randomly to either an exercise group (FCT) or a control group

Undergo Functional movement screen, endurance, jumping, and reaction time assessments before and after the 8-week period

Continue their usual fencing training throughout the study

The study will help determine whether adding corrective exercises to standard training can improve function and performance in young athletes.

DETAILED DESCRIPTION:
This randomized controlled single-blind study investigates the effects of an 8-week Functional Corrective Training (FCT) program on trunk muscle endurance, jump performance, and reaction time in adolescent fencers.

Background and Rationale:

Fencing is a dynamic sport that demands high levels of coordination, agility, strength, and cognitive processing. Due to its asymmetric and high-intensity nature, fencing may lead to movement pattern deficiencies, postural imbalances, and a higher risk of overuse injuries, particularly during adolescence-a critical period for neuromuscular development. Functional Movement Screen (FMS) is a validated tool used to identify these deficiencies, and Functional Corrective Training exercises based on FMS results aim to improve fundamental movement patterns, mobility, and stability.

While prior studies have demonstrated the positive effects of FCT on FMS scores and injury prevention, there is limited and inconsistent evidence on its impact on athletic performance. This study is the first to explore the efficacy of FCT on posture and performance in adolescent fencers, a population with unique sport-specific movement demands.

Study Design and Procedures:

Participants aged 10-19 years, with at least three years of fencing experience and no current pain or recent injury, were randomly assigned to either the FCT group or the control group. Randomization was performed using SPSS software. The intervention group received an individualized 8-week FCT program designed using the FMS Pro 360 software based on each participant's FMS results. The program progressed weekly and was applied under supervision (3 sessions/week) and as a home-based program (3 sessions/week). The control group continued their standard fencing training without additional corrective exercises.

Assessments were conducted at baseline and after the 8-week intervention by two physiotherapists blinded to group allocation. Primary outcome measures included trunk endurance (McGill tests), jump performance (CMJ and SLJ using OptoJump), and reaction time (via optical stimulus response). FMS scores were also evaluated to assess changes in movement patterns.

Data Quality and Management Procedures:

All data were entered into an anonymized electronic database and cross-verified by two independent researchers.

Range and consistency checks were applied to each entry point to ensure data validity.

Source data verification was performed for 20% of participants by comparing the collected data with original forms and digital measurements (OptoJump system output).

A data dictionary was prepared including definitions, coding methods, and measurement units for all variables.

Standard Operating Procedures (SOPs) were followed for data collection, storage, participant follow-up, and adverse event reporting.

Participants were instructed and monitored by certified physiotherapists throughout the program. Compliance with home programs was supervised by club trainers, and adherence was documented weekly.

Sample Size and Statistical Analysis:

The study began with 32 participants (n=16 per group). Following attrition, 22 participants (n=11 per group) completed the study. While no formal power analysis was conducted due to the pilot nature of the study, the sample size was deemed adequate to observe preliminary effects.

Descriptive statistics were used to summarize demographic data. Normality of data distribution was assessed using the Shapiro-Wilk test, histograms, and Q-Q plots. Between-group comparisons were made using independent samples t-test or Mann-Whitney U test depending on data distribution. Within-group changes were evaluated with paired t-tests or Wilcoxon signed-rank tests. Statistical significance was set at p < 0.05.

Handling of Missing Data:

Participants with incomplete assessments or missing post-intervention data were excluded from the final analysis. No data imputation was performed. All analyses were conducted on a per-protocol basis.

Safety and Monitoring:

No adverse events related to the intervention were reported. All exercises were performed under professional supervision, and participants were instructed to report any discomfort or issues during sessions.

This study aims to provide new insights into how individualized corrective exercise programs can enhance postural control, muscular endurance, and performance in young athletes, potentially offering a preventive and performance-enhancing strategy for youth sport training.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 10 to 19 years
* Practicing fencing for at least 3 years
* Currently pain-free in all body regions
* Able and willing to participate in regular training and assessment sessions
* Provided informed consent (and parental consent where applicable)

Exclusion Criteria:

* History of sports injury or musculoskeletal rehabilitation in the past 6 months
* Currently following a specialized exercise program other than the standard strength and conditioning routine used in the club
* Inability to commit to the full 8-week intervention period or scheduled assessments
* Any neurological, orthopedic, or systemic conditions affecting movement or physical performance

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Trunk Muscle Endurance | Baseline and 8 weeks
  Assessed using McGill's core endurance tests (flexion, extension, right and left side bridge tests) in seconds.
Change in Jump Performance | Baseline and 8 weeks
  Measured by Countermovement Jump (CMJ) and Single-Leg Jump (SLJ) height using the OptoJump system /height in centimeters

SECONDARY OUTCOMES:
Change in Reaction Time | Baseline and 8 weeks
  Measured via optical stimulus using the OptoJump system for both dominant and non-dominant legs

CONTACTS AND LOCATIONS:
Overall Officials: Seda Bicici Ulusahin, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri Universitesi, Ankara, Kecioren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to concerns regarding participant confidentiality and the lack of explicit consent for data sharing, the individual participant data will not be made available to other researchers.

REFERENCES:
- [Background] Reiman MP, Krier AD, Nelson JA, Rogers MA, Stuke ZO, Smith BS. Comparison of different trunk endurance testing methods in college-aged individuals. Int J Sports Phys Ther. 2012 Oct;7(5):533-9. PMID 23091786
- [Background] Aitken ME, Jaffe KM, DiScala C, Rivara FP. Functional outcome in children with multiple trauma without significant head injury. Arch Phys Med Rehabil. 1999 Aug;80(8):889-95. doi: 10.1016/s0003-9993(99)90079-5. PMID 10453764
- [Background] Hosseinzadeh Nik T, Shahsavari N, Ghadirian H, Ostad SN. Acetaminophen Versus Liquefied Ibuprofen for Control of Pain During Separation in Orthodontic Patients: A Randomized Triple Blinded Clinical Trial. Acta Med Iran. 2016 Jul;54(7):418-21. PMID 27424011
- [Background] Mau H, Baker RT. A modified mobilization-with-movement to treat a lateral ankle sprain. Int J Sports Phys Ther. 2014 Aug;9(4):540-8. PMID 25133082
- [Background] Pietrosimone B, Thomas AC, Saliba SA, Ingersoll CD. Association between quadriceps strength and self-reported physical activity in people with knee osteoarthritis. Int J Sports Phys Ther. 2014 May;9(3):320-8. PMID 24944850
- [Background] O'Brien W, Khodaverdi Z, Bolger L, Tarantino G, Philpott C, Neville RD. The Assessment of Functional Movement in Children and Adolescents: A Systematic Review and Meta-Analysis. Sports Med. 2022 Jan;52(1):37-53. doi: 10.1007/s40279-021-01529-3. Epub 2021 Sep 15. PMID 34524655
- [Background] Sti. Vegane Diat wirkt auch uber das Mikrobiom. MMW Fortschr Med. 2019 Oct;161(18):19. doi: 10.1007/s15006-019-0988-4. No abstract available. German. PMID 31631267
- [Background] Nishiki-Muranishi N, Harada Y, Minamikawa T, Yamaoka Y, Dai P, Yaku H, Takamatsu T. Label-free evaluation of myocardial infarction and its repair by spontaneous Raman spectroscopy. Anal Chem. 2014 Jul 15;86(14):6903-10. doi: 10.1021/ac500592y. Epub 2014 Jun 23. PMID 24914734
- [Background] Howatson G, van Someren KA. The prevention and treatment of exercise-induced muscle damage. Sports Med. 2008;38(6):483-503. doi: 10.2165/00007256-200838060-00004. PMID 18489195